CLINICAL TRIAL: NCT03563755
Title: Social Information Processing in Adolescents With Eating Disorders: Implications for Theory and Clinical Practice
Brief Title: Social Information Processing in Adolescents With Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); South West London and St George's Mental Health NHS Trust (Other); Ellern Mede Ridgeway (Unknown); Ellern Mede Barnet (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 229005
Record Dates: First submitted 2018-05-09; First posted 2018-06-20 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Eating Disorders in Adolescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification (CBM) + Treatment as usual (Experimental): Participants will receive access to a 3-week online training programme alongside their usual treatment.
  Interventions: Other: Cognitive Bias Modification
- Treatment as usual (No Intervention): Participants will continue to receive their usual treatment.

INTERVENTIONS:
Other: Cognitive Bias Modification — CBM-Attention (CBM-A) will be used with the aim of ameliorating negative cognitive biases in attention by redirecting attention towards positive social stimuli (accepting faces). Similarly CBM-Interpretation (CBM-I) will be used to ameliorate negative interpretation bias, by reinforcing benign outcomes of ambiguous social scenarios. Implementation intentions will be used to guide participants in planning new ways to face difficult social situations involving the risk of social rejection/criticism. Participants will continue to receive their usual treatment.
  Arms: Cognitive Bias Modification (CBM) + Treatment as usual

SUMMARY:
This research project aims to examine whether adding an online programme of cognitive training exercises may be a helpful addition to treatment as usual for young people with eating disorders. The cognitive training exercises aim to modify distortions in attention and thinking during hypothetical, ambiguous social interactions involving the risk of social rejection.

All participants will complete a baseline assessment consisting of a battery of questionnaires and computerised tasks, to assess attention and thinking during ambiguous social interactions involving the risk of social rejection. Participants who display distortions in attention and thinking will then be randomised to one of two groups. In one group participants will receive the computerised training alongside their usual treatment. In the other group participants will continue to receive their treatment as usually only.

Healthy controls will also be invited to take part in the baseline assessment to allow for comparisons between clinical and non-clinical groups.

DETAILED DESCRIPTION:
The aim of this study is to assess the effects of adding 10 sessions of Cognitive Bias Modification (CBM) training, and goal planning using implementation intentions, to treatment as usual for adolescents with eating disorders. It is hypothesised that at baseline, participants will demonstrate cognitive biases in their attention towards rejecting/critical facial expressions (attentional bias), and in making negative resolutions of ambiguous social scenarios involving the risk of social rejection (interpretation bias).

Young people receiving treatment for eating disorders will be recruited from participating child and adolescent eating disorder services in the United Kingdom. Information about the study, the main eligibility criteria and contact details for the researcher will also be advertised using flyers and social media platforms. Individuals from the community who express an interest in taking part will be screened using the Structured Clinical Interview for DSM-5 (SCID-5) disorders to screen for psychiatric disorders to determine their eligibility. Parental consent will be obtained for any participants under the age of 16. Eligible participants will be invited to meet the researcher for an initial visit, to provide consent and complete the baseline assessments. The baseline assessments will consist of a battery of questionnaires used to assess interpersonal sensitivity, mood, anxiety and eating disorder psychopathology, and computerised tasks to measure various aspects of social cognition including attention and interpretation biases.

Following the baseline assessments, participants displaying attention and interpretation biases will be invited to take part in the next phase of the study. Participants randomised to receive the computerised training will meet with the researcher for a second visit, during which they will learn how to complete the training tasks, complete the first set of training modules and create plans involving exposure to the risk of social rejection with the researcher using the implementation intentions approach. Participants will be asked to complete the remaining training three times per week over three weeks (10 sessions in total) and will have weekly contact with the researcher to review adherence to planned behaviours using implementations intentions. Attention and interpretation biases will be assessed again at the end of the 3-week training and at 12 weeks follow-up. Questionnaire measures of interpersonal sensitivity, anxiety, depression and disorder psychopathology will also be administered at these two time points.

ELIGIBILITY:
Inclusion Criteria for patients with eating disorders

* Fluency in English
* Aged 13-17
* With an eating disorder diagnosis according to the DSM-5

Exclusion Criteria:

* Severe psychiatric comorbidity requiring treatment in its' own right (e.g. psychosis)
* Neurological condition (e.g. epilepsy)
* Severe visual impairment uncorrected with visual aids (eyewear)
* Not receiving specialist treatment for an eating disorder

Inclusion Criteria for healthy volunteers

* Fluency in English
* Aged 13-17

Exclusion Criteria:

* Current psychiatric diagnosis according to the DSM-5 (e.g. depression, anxiety)
* History of a psychiatric disorder
* Neurological condition (e.g. epilepsy)
* Severe visual impairment uncorrected with visual aids (eyewear)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-03-28 (Estimated); Study Completion 2020-03-28 (Estimated)

PRIMARY OUTCOMES:
Change in attentional bias towards positively valenced faces | End of intervention (3 weeks post-randomisation)
  Attentional probe assessment task and visual search task: reaction times (milliseconds) and accuracy
Change in positive interpretations of ambiguous social scenarios | End of intervention (3 weeks post-randomisation)
  Sentence completion task and test trials from ambiguous scenarios training (frequencies of positive, neutral and negative interpretations).

SECONDARY OUTCOMES:
Change in self-reported frequency of experiencing various symptoms of anxiety | End of intervention (3 weeks post-randomisation)
  Score on the Revised Child Anxiety and Depression Scale (RCADS). A higher score reflects a greater degree of symptom severity. Converted scores on the total scale and both sub-scales are divided into three scoring ranges, 1) Scores below 65 represent low severity 2) Scores between 65-70 represent medium severity and are on the borderline clinical threshold 3) Scores above 70 represent high severity and are above the clinical threshold.
Change in self-reported frequency of experiencing various symptoms of low mood | End of intervention (3 weeks post-randomisation)
  Score on the Revised Child Anxiety and Depression Scale (RCADS). A higher score reflects a greater degree of symptom severity. Converted scores on the total scale and both sub-scales are divided into three scoring ranges, 1) Scores below 65 represent low severity 2) Scores between 65-70 represent medium severity and are on the borderline clinical threshold 3) Scores above 70 represent high severity and are above the clinical threshold.
Change in Eating Disorder symptoms | End of intervention (3 weeks post-randomisation)
  Scores on the Eating Disorder Examination Questionnaire (EDE-Q). The EDE-Q is scored using a 7-point, forced-choice rating scale (0-6) with scores of 4 or higher indicative of clinical range. Subscale and global scores reflect the severity of eating disorder psychopathology. To obtain subscale scores, the ratings for the relevant items are added together and the sum is then divided by the total number of items forming the subscale. A "global" score is the sum of the four subscale scores divided by the number of subscales (i.e., four).
Change in self-reported interpersonal sensitivity | End of intervention (3 weeks post-randomisation)
  Scores on the Interpersonal Sensitivity Measure (IPSM). The IPSM is a 36-item measure. Each item is rated on a four-point scale, ranging from 4 (very like me) to 1 (very unlike me), with higher scores reflecting greater concerns about experiences involving the risk of social rejection. The scale generates a total score ranging from 36 to 144.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Cardi, PhD, Study Director — King's College London
Locations (1):
- King's College London, London, United Kingdom